CLINICAL TRIAL: NCT02988973
Title: A Phase 3 Multi-center, Randomized, Open-label, Active-comparator (Darbepoetin Alfa) Conversion Study of Intermittent Oral Dosing of ASP1517 in Non-dialysis Chronic Kidney Disease Patients With Anemia
Brief Title: A Study of Intermittent Oral Dosing of ASP1517 in Non-Dialysis Chronic Kidney Disease Patients With Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Kyntra Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1517-CL-0310
Record Dates: First submitted 2016-12-08; First posted 2016-12-12 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Chronic Kidney Disease
Keywords: Roxadustat; Anemia; Non-dialysis chronic kidney disease; ASP1517
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia | interventions — roxadustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- rHuEPO or DA to ASP1517 (Experimental): Participants will receive roxadustat according to the prior randomization treatment, with starting doses of 70mg thrice weekly (TIW) to participants on <4500 IU/week of rHuEPO or <20 microgram (μg)/week of darbepoetin alfa (DA) and 100mg TIW to participants on ≥4500 IU/week rHuEPO or ≥ 20 μg/week DA. Participants roxadustat dosage will be adjusted every 4 weeks to maintain Hb level within the target range 10.0 to 12.0 g/dL. Dose adjustment steps will be as follows: 20, 40, 50, 70, 100, 150, 200, 250, 300 mg.
  Interventions: Drug: roxadustat
- rHuEPO or DA to DA (Experimental): Participants will receive DA according to the prior randomization treatment, with starting doses of 15 μg/2weeks to participants on ≤ 1500 IU/week of rHuEPO or <11.25 microgram (μg)/week of DA, 30μg/2weeks to participants on >1500 to <6000 IU/week of rHuEPO or ≥ 11.25 to < 22.5 μg/week of DA, 60μg/2weeks to participants on ≥ 6000 IU/week of rHuEPO or ≥ 22.5 to < 37.5 μg/week of DA, 90μg/2weeks to participants on ≥ 37.5 to < 52.5 μg/week of DA, 120μg/2weeks to participants on ≥ 52.5 to < 75 μg/week of DA, 180μg/2weeks to participants on ≥ 75 μg/week of DA. Participant's roxadustat dosage will be adjusted every 4 weeks to maintain Hb level within the target range 10.0 to 12.0 g/dL. Dose adjustment steps will be as follows: 15, 30, 60, 90, 120, and 180 μg.
  Interventions: Drug: DA
- Epoetin beta pegol to ASP1517 (Experimental): Participants will receive roxadustat according to the prior registration treatment, with starting doses of 70mg thrice weekly (TIW) to participants on ≤100 μg/week of Epoetin beta pegol and 100mg TIW to participants on >100 μg/week of Epoetin beta pegol. Participant's roxadustat dosage will be adjusted every 4 weeks to maintain Hb level within the target range 10.0 to 12.0 g/dL. Dose adjustment steps will be as follows: 20, 40, 50, 70, 100, 150, 200, 250, 300 mg.
  Interventions: Drug: roxadustat

INTERVENTIONS:
Drug: roxadustat — Oral administration
  Other Names: ASP1517
  Arms: Epoetin beta pegol to ASP1517; rHuEPO or DA to ASP1517
Drug: DA — Subcutaneous administration
  Arms: rHuEPO or DA to DA

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of ASP1517 when converted from recombinant human erythropoietin (rHuEPO) or darbepoetin alfa (DA), compared to DA in the treatment of anemia in non-dialysis chronic kidney disease patients. Another uncontrolled cohort will be included to evaluate the efficacy and safety of ASP1517 in patients converted from epoetin beta pegol (CERA). This study will also assess the safety/efficacy of long term treatment of ASP1517 (52 weeks).

DETAILED DESCRIPTION:
This study consists of the following three cohorts. Cohort 1; subjects converted from rHuEPO or DA to ASP1517, Cohort 2; subjects converted from rHuEPO or DA to DA, Cohort 3; subjects converted from epoetin beta pegol (CERA) to ASP1517. In Cohort 1 and 3, ASP1517 will be administered orally for 52 weeks. In Cohort 2, DA will be administered subcutaneously for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who were diagnosed with non-dialysis Chronic Kidney Disease and who are considered not to require renal replacement therapy during the study period
* Subjects with renal anemia who have been receiving erythropoiesis stimulating agent (ESA) by subcutaneous injection and whose Hb values are considered stable.
* Mean of the subject's two most recent Hb values before randomization during the Screening Period must be ≥10.0 g/dL and ≤12.0 g/dL
* Either transferrin saturation ≥ 20% or serum ferritin ≥ 100 ng/mL
* Female subject must either:

Be of non-childbearing potential:

* post-menopausal, or
* documented surgically sterile Or, if of childbearing potential,
* Agree not to try to become pregnant during the study and for 28 days after the final study drug administration
* And have a negative urine pregnancy test at pre-screening
* And, if heterosexually active, agree to consistently use two forms of highly effective birth control* (at least one of which must be a barrier method) starting at pre-screening and throughout the study period and continued for 28 days after the final study drug administration.

  * Female subject must agree not to breastfeed starting at pre-screening and throughout the study period, and continued for 28 days after the final study drug administration.
  * Female subject must not donate ova starting at pre-screening and throughout the study period, and continued for 28 days after the final study drug administration.
  * Male subject and their female spouse/partners who are of childbearing potential must be using two forms of highly effective birth control (at least one of which must be a barrier method) starting at pre-screening and continue throughout the study period, and for 12 weeks after the final study drug administration
  * Male subject must not donate sperm starting at pre-screening and throughout the study period and, for 12 weeks after the final study drug administration

Exclusion Criteria:

* Concurrent retinal neovascular lesion untreated or macular edema untreated, and patients with any condition that significantly compromises the ability to visualize the retina
* Concurrent autoimmune disease with inflammation that could impact erythropoiesis
* History of gastric/intestinal resection considered influential on the absorption of drugs in the gastrointestinal tract (excluding resection of gastric or colon polyps) or concurrent gastro-paresis
* Uncontrolled hypertension
* Concurrent congestive heart failure (NYHA Class III or higher)
* History of hospitalization for treatment of stroke, myocardial infarction, or pulmonary embolism within 12 weeks before the pre-screening assessment
* Positive for hepatitis B surface antigen (HBsAg) or anti-hepatitis C virus (HCV) antibody at the pre-screening assessment, or positive for human immunodeficiency virus (HIV) in a past test
* Concurrent other form of anemia than renal anemia
* History of pure red cell aplasia
* Having received treatment with protein anabolic hormone, testosterone enanthate, or mepitiostane within 6 weeks before the pre-screening assessment
* Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), or total bilirubin that is greater than the criteria, or previous or concurrent another serious liver disease at pre-screening assessment
* Previous or current malignant tumor (no recurrence for at least 5 years is eligible.)
* Having undergone red blood transfusion and/or a surgical procedure consider to promote anemia and/or ophthalmological surgery within 4 weeks before the pre-screening assessment
* Having undergone a kidney transplantation
* History of serious drug allergy including anaphylactic shock
* Having a previous history of treatment with ASP1517 or participation in this study
* Participation in another clinical study or post-marketing clinical study (including that of a medical device) within 12 weeks before informed consent acquisition

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2019-09-13 (Actual); Study Completion 2020-03-26 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the average Hemoglobin (Hb) | Baseline and Weeks 18 to 24

SECONDARY OUTCOMES:
Average Hb from Week 18 to Week 24 | Up to Week 24
Number of Participants Who Achieved the Average Hb level of 10.0 to 12.0 g/dL For Weeks 18 to 24 | Weeks 18 to 24
Number of participants who achieve the target Hb level at each week | Up to Week 24
Change from baseline in Hb to each post-dosing time point | Baseline and Up to Week 52
Proportion of time points that achieve the target Hb level from Weeks 18 to 24 | Up to Week 24
Rate of rise in Hb levels (g/dL/week) from week 0 to at the earliest date of week 4, time of discontinuation, or time of dose adjustment | Up to Week 4
Quality of life assessed by SF-36 | Up to Week 52
  SF-36: Medical Outcomes Study 36-Item Short-Form Health Survey
Quality of life assessed by EQ-5D-5L | Up to Week 52
  EQ-5D: EuroQol 5 Dimension 5 Levels
Quality of life assessed by WPAI:ANS | Up to Week 52
  WPAI:ANS: Work Productivity and Activity Impairment Questionnaire: Anaemic Symptoms
Quality of life assessed by FACT-An | Up to Week 52
  FACT-An: Functional Assessment of Cancer Therapy-Anemia
Average Hb from weeks 44 to 52 | Up to Week 52
Change from baseline in the average Hb from weeks 44 to 52 | Baseline and Up to Week 52
Number of Participants Who Achieved the Average Hb level of 10.0 to 12.0 g/dL For Weeks 44 to 52 | Weeks 44 to 52
Number of participants who achieve the target Hb level at each week | Up to Week 52
Proportion of time points that achieve the target Hb level from Weeks 44 to 52 | Up to Week 52
Average Hematocrit Level | Up to Week 52
Average Reticulocyte Level | Up to Week 52
Average Ferrum Level | Up to Week 52
Average Ferritin Level | Up to Week 52
Average Transferrin Level | Up to Week 52
Average Total Iron Binding Capacity Level | Up to Week 52
Average Soluble Transferrin Receptor Level | Up to Week 52
Average Soluble Transferrin Level | Up to Week 52
Average Reticulocyte Hemoglobin Content Level | Up to Week 52
Number of Occurence of Hospitalizations | Up to Week 52
Duration of Hospitalization | Up to week 52
Number of participants with abnormal Vital signs and/or adverse events related to treatment | Up to Week 52
Safety assessed by body weight | Up to Week 52
Safety assessed by incidence of adverse events | Up to Week 52
Safety assessed by standard 12-lead electrocardiogram | Up to Week 52
Safety assessed by ophthalmological examination: Fundoscopy | Up to Week 24
Safety assessed by ophthalmological examination: optical coherence tomography | Up to Week 24
Safety assessed by ophthalmological examination: visual acuity | Up to Week 24
Number of participants with abnormal Laboratory values and/or adverse events related to treatment | Up to Week 52
Plasma concentration of unchanged ASP1517 | Up to Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (66):
- Japan (66):
  - Site JP00009, Kasugai, Aichi-ken
  - Site JP00030, Nagoya, Aichi-ken
  - Site JP00051, Nagoya, Aichi-ken
  - Site JP00021, Toyohashi, Aichi-ken
  - Site JP00003, Sakura, Chiba
  - Site JP00038, Matsuyama, Ehime
  - Site JP00044, Matsuyama, Ehime
  - Site JP00008, Kitakyushu, Fukuoka
  - Site JP00013, Kitakyushu, Fukuoka
  - Site JP00040, Kitakyushu, Fukuoka
  - Site JP00057, Kitakyushu, Fukuoka
  - Site JP00042, Kurume, Fukuoka
  - Site JP00041, Tajimi, Gifu
  - Site JP00002, Maebashi, Gunma
  - Site JP00037, Hatsukaichi, Hiroshima
  - Site JP00050, Kure, Hiroshima
  - Site JP00049, Aasahikawa, Hokkaido
  - Site JP00007, Sapporo, Hokkaido
  - Site JP00064, Sapporo, Hokkaido
  - Site JP00022, Amagasaki, Hyōgo
  - Site JP00066, Nishinomiya, Hyōgo
  - Site JP00052, Hitachi, Ibaraki
  - Site JP00017, Kasama, Ibaraki
  - Site JP00028, Koga, Ibaraki
  - Site JP00053, Naka, Ibaraki
  - Site JP00023, Sashima-gun, Ibaraki
  - Site JP00019, Toride, Ibaraki
  - Site JP00046, Tsuchiura, Ibaraki
  - Site JP00035, Kanazawa, Ishikawa-ken
  - Site JP00031, Morioka, Iwate
  - Site JP00047, Fujisawa, Kanagawa
  - Site JP00001, Kamakura, Kanagawa
  - Site JP00016, Yokohama, Kanagawa
  - Site JP00048, Yokohama, Kanagawa
  - Site JP00012, Sendai, Miyagi
  - Site JP00036, Ueda, Nagano
  - Site JP00059, Higashiosaka, Osaka
  - Site JP00005, Izumisano, Osaka
  - Site JP00011, Sakai, Osaka
  - Site JP00069, Yao, Osaka
  - Site JP00029, Ageo, Saitama
  - Site JP00004, Koshigaya, Saitama
  - Site JP00020, Koshigaya, Saitama
  - Site JP00025, Adachi-ku, Tokyo
  - Site JP00043, Bunkyo-ku, Tokyo
  - Site JP00063, Chiyoda-ku, Tokyo
  - Site JP00067, Hino, Tokyo
  - Site JP00015, Koto-ku, Tokyo
  - Site JP00024, Minato-ku, Tokyo
  - Site JP00006, Musashino, Tokyo
  - Site JP00060, Ōta-ku, Tokyo
  - Site JP00062, Tachikawa, Tokyo
  - Site JP00014, Fukui
  - Site JP00033, Fukuoka
  - Site JP00065, Fukuoka
  - Site JP00032, Hiroshima
  - Site JP00039, Hiroshima
  - Site JP00045, Kyoto
  - Site JP00018, Nagano
  - Site JP00068, Nagano
  - Site JP00026, Niigata
  - Site JP00055, Okayama
  - Site JP00056, Osaka
  - Site JP00061, Osaka
  - Site JP00034, Ōita
  - Site JP00010, Toyama

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278
- [Derived] Akizawa T, Tanaka-Amino K, Otsuka T, Yamaguchi Y. Factors Affecting Doses of Roxadustat Versus Darbepoetin Alfa for Anemia in Nondialysis Patients. Am J Nephrol. 2021;52(9):702-713. doi: 10.1159/000519043. Epub 2021 Oct 8. PMID 34628408
- See also: Link to results on the Astellas Clinical Study. — https://astellasclinicalstudyresults.com/hcp/study.aspx?ID=398